CLINICAL TRIAL: NCT01316588
Title: Recolonization of the Skin Following Pre-operative Disinfection and Impact of the Use of Plastic Adhesive Drapes
Brief Title: Recolonization Following Preoperative Disinfection Plastic Adhesive Drapes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Örebro University, Sweden (Other)
Collaborators: Region Örebro County (Other)
Responsible Party: Principal Investigator, Ulrica Nilsson, Professor, Örebro University, Sweden
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2010/46
Record Dates: First submitted 2011-03-11; First posted 2011-03-16 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Surgical Wound Infection
Keywords: recolonization; Plastic adhesive drape; microbial sealant; SSI; bacterial growth
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Plastic adesive drape (Experimental): Intraoperative: Plastic adhesive drape on the chest and bare skin on the leg
  Interventions: Other: Plastic adesive drape
- Microbial Sealant (Experimental): Intraoperative: Microbial Sealant on the leg and bare skin on the chest
  Interventions: Other: Microbial Sealant

INTERVENTIONS:
Other: Plastic adesive drape — Plastic adhesive drape intraoperatively on patients skin around the surgical wound on the chest and bare skin on the leg
  Arms: Plastic adesive drape
Other: Microbial Sealant — Microbial sealant intraoperatively on patients skin around the surgical wound on the leg and bare skin on the chest
  Arms: Microbial Sealant

SUMMARY:
The purpose of this study is to measure the time to recolonization intraoperatively after preoperative disinfection with chlorhexidine solution in ethanol and to determine evidence of differential bacterial growth with or without plastic adhesive drape on the chest as well as with or without microbial sealant on the leg.

DETAILED DESCRIPTION:
The purpose of this study is to measure the time to recolonization intraoperative after preoperative disinfection with chlorhexidine solution in ethanol and to determine evidence of differential bacterial growth with or without plastic adhesive drape as well as with or without microbial sealant on the leg. A RCT study of 140 patients undergoing coronary artery bypass grafting (CABG) and/or aortic valve replacement (AVR) are included. The investigators test the hypothesis that patients randomized to no plastic adhesive drape intraoperatively will have a reduced recolonisation compared to patients with plastic adhesive drape.

ELIGIBILITY:
Inclusion Criteria:

Elective CABG and/or AVR

Exclusion Criteria:

Suffer from any recent infection two weeks prior to the start of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2010-08; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Bacterial samples | Bacterial samples are taken on eight occasionson the chest and at five occations
  Bacterial samples on the skin of the chest: one day before surgery, the day of surgery, and immediately after disinfection. Thereafter five times both on the skin and in the surgical wound i.e. 60, 120, 180 and 240 minutes intraoperatively as well as at the closure of the surgical wound.
  Bacterial samples on the leg: one day before surgery, the day of surgery, and immediately after disinfection. Thereafter at two occasions both : on the skin and in the surgical wound i.e. at the incision and at the closure of the surgical wound.

SECONDARY OUTCOMES:
Surgical site infection | once
  ASEPSIS score will be measured after 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Ulrica Nilsson, PhD, Professor, Principal Investigator — Örebro University, faculty of Medicine and Health , Sweden
Locations (1):
- Orebro University, Faculty of medicine and Health, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Falk-Brynhildsen K, Soderquist B, Friberg O, Nilsson U. Bacterial growth and wound infection following saphenous vein harvesting in cardiac surgery: a randomized controlled trial of the impact of microbial skin sealant. Eur J Clin Microbiol Infect Dis. 2014 Nov;33(11):1981-7. doi: 10.1007/s10096-014-2168-x. Epub 2014 Jun 8. PMID 24907853
- [Result] Falk-Brynhildsen K, Soderquist B, Friberg O, Nilsson UG. Response to M.H. Stevens and N.M. Klinger, re: Bacterial recolonization of the skin and wound contamination during cardiac surgery. J Hosp Infect. 2013 Dec;85(4):325. doi: 10.1016/j.jhin.2013.09.001. Epub 2013 Sep 17. No abstract available. PMID 24080082
- [Result] Falk-Brynhildsen K, Soderquist B, Friberg O, Nilsson UG. Bacterial recolonization of the skin and wound contamination during cardiac surgery: a randomized controlled trial of the use of plastic adhesive drape compared with bare skin. J Hosp Infect. 2013 Jun;84(2):151-8. doi: 10.1016/j.jhin.2013.02.011. Epub 2013 Apr 25. PMID 23623487